CLINICAL TRIAL: NCT01507233
Title: A Pain Relief Trial Utilizing the Infiltration of a Multivesicular Liposome Formulation Of Bupivacaine, EXPAREL®: A Phase 4 Health Economic Trial in Adult Patients Undergoing Open Colectomy
Brief Title: A Health Economic Trial in Adult Patients Undergoing Open Colectomy MA402S23B302
Acronym: IMPROVE-Open
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MA402S23B302
Record Dates: First submitted 2011-10-24; First posted 2012-01-10 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-01

CONDITIONS: Bowel Obstruction
Keywords: open colectomy; colectomy
MeSH Terms: conditions — Intestinal Obstruction | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV morphine sulfate (Active Comparator): morphine sulfate (or Sponsor-approved equivalent)
  Interventions: Drug: IV morphine sulfate
- EXPAREL (Experimental): EXPAREL (bupivacaine liposome injectable suspension)
  Interventions: Drug: EXPAREL (bupivacaine liposome injectable suspension)

INTERVENTIONS:
Drug: IV morphine sulfate — Patients in this group will receive IV morphine sulfate via patient-controlled analgesia (PCA) pump, as needed. The PCA pump will be set up postsurgically as soon as possible and prior to the patient leaving the post-anesthesia care unit (PACU) or immediately upon transfer to the floor if the stay in the PACU is less than 1 hour.
  Other Names: morphine sulfate (or Sponsor-approved equivalent)
  Arms: IV morphine sulfate
Drug: EXPAREL (bupivacaine liposome injectable suspension) — Patients in this group will receive 266 mg EXPAREL diluted with preservative free 0.9% normal saline to a total volume of 30 cc and administered via wound infiltration prior to wound closure. When not contraindicated, 30 mg IV ketorolac, a non-steroidal anti-inflammatory drug (NSAID), may be substituted per the site's standard of care.
  All patients will be offered rescue analgesia, as needed.
  Other Names: bupivacaine free base
  Arms: EXPAREL

SUMMARY:
This study is designed to compare the standard of care against EXPAREL (bupivacaine liposome extended-release injectable suspension) to determine if total opioid consumption is reduced when using EXPAREL, therefore possibly reducing total hospitalization costs.

DETAILED DESCRIPTION:
This is a phase 4, prospective, sequential, open-label study designed to evaluate the efficacy, safety, and health economic benefits of intraoperative local wound infiltration with EXPAREL (bupivacaine liposome extended-release injectable suspension), compared with postsurgical administration of standardized intravenous (IV) morphine sulfate, for postsurgical analgesia in adult patients undergoing open colectomy with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Patients scheduled to undergo open segmental colectomy with planned primary anastamosis, as defined by cecectomy, right hemicolectomy, resection of transverse colon, left hemicolectomy, or sigmoidectomy.
* Ability to provide informed consent, adhere to study visit schedule, and complete all assessments.

Exclusion Criteria:

* Patients with a history of hypersensitivity or idiosyncratic reactions or intolerance to any local anesthetic, opioid, or propofol.
* Patients who abuse alcohol or other drug substance.
* Patients with severe hepatic impairment.
* Patients currently pregnant or who may become pregnant during the course of the study.
* Patients with any psychiatric, psychological, or other condition that the Investigator feels may make the patient an inappropriate candidate for this clinical study.
* Patients who have participated in a EXPAREL study within the last 30 days.
* Patients who have received an investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the patient's participation in this study.
* Patients who undergo any concurrent surgical procedure during the ileostomy reversal surgery.

In addition, the patient will be ineligible if he/she meets the following criteria during surgery:

* Patients with unplanned multiple segmental resections or large intestine.
* Patients who have unplanned, temporary or permanent colostomies, ileostomies, or the like placed.
* Patients who receive intraoperative administration of opioids (other than fentanyl or analogs) or an other analgesic, local anesthetics, or anti-inflammatory agents.
* Patients who receive Entereg(R).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Candiotti, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Dept of Anesthesiology, Miami, Florida, United States

REFERENCES:
- [Derived] Cohen SM, Vogel JD, Marcet JE, Candiotti KA. Liposome bupivacaine for improvement in economic outcomes and opioid burden in GI surgery: IMPROVE Study pooled analysis. J Pain Res. 2014 Jun 24;7:359-66. doi: 10.2147/JPR.S63764. eCollection 2014. PMID 25018650

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Morphine Sulfate: morphine sulfate (or Sponsor-approved equivalent)
  IV morphine sulfate: Patients in this group will receive IV morphine sulfate via PCA pump, as needed. The PCA pump will be set up postsurgically as soon as possible and prior to the patient leaving the PACU or immediately upon transfer to the floor if the stay in the PACU is less than one hour.
- EXPAREL: EXPAREL (bupivacaine liposome injectable suspension)
  EXPAREL (bupivacaine liposome injectable suspension): Patients in this group will receive 266 mg EXPAREL diluted with preservative free 0.9% normal saline to a total volume of 30 cc and administered via wound infiltration prior to wound closure. When not contraindicated, 30 mg IV ketorolac, a non-steroidal anti-inflammatory drug (NSAID), may be substituted per the site's standard of care.
  All patients will be offered rescue analgesia, as needed.
Period: Overall Study
Arm/Group | IV Morphine Sulfate | EXPAREL
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Morphine Sulfate | EXPAREL | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.76) |  | 53.6 (13.76)
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 4 |  | 4
  >=65 years | 1 |  | 1
Gender [Number; unit: participants]
  Female | 3 |  | 3
  Male | 2 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Burden
Description: Total opioid consumed (IV and PO) postsurgically until the hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order written or Day 30, whichever is sooner
Population: As no subjects received EXPAREL in this study, statistical analyses were not performed.
Arm/Group | IV Morphine Sulfate | EXPAREL
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Health Economic Benefits
Description: 1. Total cost of hospitalization until the time hospital discharge order is written or through Day 30, whichever is sooner.
  2. Length of stay (LOS), recorded in hours, defined as the time of completion of the wound closure until the hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to Day 30
Population: As no subjects received EXPAREL in this study, statistical analyses were not performed.
Arm/Group | IV Morphine Sulfate | EXPAREL
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Opioid-related Adverse Events and Patient Satisfaction With Postsurgical Analgesia.
Description: 1. Incidence of opioid-related adverse events defined as somnolence, respiratory depression, hypoventilation, hypoxia, dry mouth, nausea, vomiting, constipation, sedation, confusion, pruritus, urinary retention, and postoperative ileus.
  2. Responses to one question pertaining to patient satisfaction with postsurgical analgesia and four questions pertaining to postsurgical recovery following hospital discharge.
Time Frame: Wound closure to time hospital discharge order written or Day 30, whichever is sooner.
Population: As no subjects received EXPAREL in this study, statistical analyses were not performed.
Arm/Group | IV Morphine Sulfate | EXPAREL
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days post surgery
Description: normal systematic assessment of adverse events
Arm/Group | IV Morphine Sulfate | EXPAREL
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Morphine Sulfate (N=5) | EXPAREL (N=0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Morphine Sulfate (N=5) | EXPAREL (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Urine output decreased (Investigations) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anemia post-operative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No